CLINICAL TRIAL: NCT06672523
Title: A Phase 1 Study to Evaluate the Mass Balance, Metabolism, Excretion, and Pharmacokinetics of [14C]-BMS-986504 (MRTX1719) in Patients With Advanced Solid Tumors With Homozygous MTAP Deletion
Brief Title: A Study to Evaluate the Mass Balance, Metabolism, Elimination, and Drug Levels of [14C]-BMS-986504 (MRTX1719) in Participants With Advanced Solid Tumors With Homozygous Methylthioadenosine Phosphorylase Deletion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA240-0008
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors With Homozygous MTAP Deletion
Keywords: Protein arginine methyltransferase (PRMT5); Methylthioadenosine-cooperative PRMT5 inhibitor; Homozygous methylthioadenosine phosphorylase (MTAP) deletion; Mass balance study; Metabolism; Elimination; Drug absorption; Distribution; Excretion; Radiolabeled; Absorption, distribution, metabolism, and excretion (ADME)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-BMS-986504 followed by BMS-986504 Monotherapy (Experimental): Part A: Participants will receive a single oral dose of radiolabeled [14C]-BMS-986504 on C1D1.
  Part B: Participants will receive non-radiolabeled BMS-986504, starting from C1D1 and until criteria for treatment discontinuation are met.
  Interventions: Drug: BMS-986504; Drug: [14C]-BMS-986504

INTERVENTIONS:
Drug: BMS-986504 — Specified dose on specified days
Drug: [14C]-BMS-986504 — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the mass balance, metabolism, elimination, and drug levels of [14C]-BMS-986504 (MRTX1719) in participants with advanced solid tumors with homozygous methylthioadenosine phosphorylase deletion.

ELIGIBILITY:
Inclusion Criteria

* Participants must have an advanced, unresectable, or metastatic solid tumor malignancy with a deletion of the methylthioadenosine phosphorylase (MTAP) gene.
* Participants must have received, be refractory to, be ineligible for, or be intolerant of available standard care for their cancer.

Exclusion Criteria

* Participants must not have a history of any surgical or medical conditions possibly affecting how the study drug is distributed, broken down (metabolized) and removed (excreted or eliminated) from the body.
* Participants must not have participated in a clinical study involving a radiolabeled study drug within 12 months prior to admission to the research center.
* Participants must not have a current or recent (within 3 months of study drug administration) gastrointestinal disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 2 weeks
Time of maximum observed drug concentration (Tmax) | Up to 2 weeks
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Up to 2 weeks
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to 2 weeks
Terminal elimination half-life (T-HALF) | Up to 2 weeks
Apparent total body clearance (CLT/F) | Up to 2 weeks
Apparent volume of distribution during the terminal phase (Vz/F) | Up to 2 weeks
Percentage of estimated part for the calculation of AUC(INF) (%AUC(INF)) | Up to 2 weeks
Blood-to-plasma total radioactivity (TRA) ratio | Up to 2 weeks
Total amount of administered dose recovered in urine (UR) | Up to 2 weeks
Percent of administered dose recovered in urine (%UR) | Up to 2 weeks
Renal clearance (CLR) in urine | Up to 2 weeks
Total radioactivity in UR | Up to 2 weeks
Total radioactivity in %UR | Up to 2 weeks
Total radioactivity in total amount of administered dose recovered in feces (FR) | Up to 2 weeks
Total radioactivity in percent of administered dose recovered in feces (%FR) | Up to 2 weeks
Total amount of radioactivity recovered (Rtotal) | Up to 2 weeks
Total percent of radioactivity recovered (%TOTAL) | Up to 2 weeks
TRA amount recovered and fraction of the radioactive dose in vomit if applicable | Up to 2 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 2 years
Number of participants with serious adverse events (SAEs) | Up to 2 years
Number of participants with AEs leading to discontinuation | Up to 2 years
Number of participants with drug-related AEs | Up to 2 years
Number of participants with laboratory abnormalities | Up to 2 years
Number of deaths | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON / PRA Magyarország Kft. Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html